CLINICAL TRIAL: NCT06017778
Title: Impact Of Whole Body Vibration on Planter /Dorsi Flexor Ratio, Pain and Functional Activities in Patellofemoral Pain Syndrome: Randomized Controlled Trial
Brief Title: Impact Of Whole Body Vibration on Planter /Dorsi Flexor Ratio, Pain and Functional Activities in Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa T. Elshorbagy, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004572
Record Dates: First submitted 2023-08-19; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; vibration; Planter/Dorsi ratio; pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body viberation group (Experimental)
  Interventions: Device: whole body vibration; Other: traditional exercise group
- control group (Active Comparator)
  Interventions: Other: traditional exercise group

INTERVENTIONS:
Device: whole body vibration — patients will receive WBV training in addition to traditional training will be performed on a tri-planar (mostly vertical, Z axis) oscillating vibration platform (Power PlateR pro5™; Power Plate North America, Inc., Northbrook, IL,USA) for 20-30 minutes per session. WBV training will be supervised and performed in a clinic three days a week with at least one day between each session for four weeks (total of 12 sessions).
  Arms: whole body viberation group
Other: traditional exercise group — 10 minutes warm-up (lower extremity stretching exercises), 20-30 minutes period of strength exercises with three sets of 10-15 repetitions (isometric quadriceps setting, knee extensions, double-legged wall squat), and 5 minutes cool-down (lower extremity stretching exercises). Lower extremity stretching exercises consisted of quadriceps, hamstring, gastrocnemius and iliotibial band stretching with 3 repetitions for 30 s each muscle.

SUMMARY:
Patellofemoral pain syndrome (PFPS) can significantly affect an individual's ability perform to functional activities, such as walking, running, climbing stairs, and sitting for prolonged periods.

PFPS is often associated with pain and discomfort in the front of the knee, which can limit an individual's range of motion and cause difficulty with weight-bearing activities. The pain may also be exacerbated by activities that involve bending the knee, such as squatting or kneeling.

Whole body vibration (WBV) has been suggested as a potential intervention for patellofemoral pain syndrome (PFPS). Some studies have shown that WBV can improve muscle strength, balance, and proprioception, which are all factors that may contribute to PFPS. Additionally, WBV may help reduce pain and improve functional abilities in individuals with PFPS However, the evidence for the effectiveness of WBV as an intervention for PFPS is still limited, and more research is needed to fully understand its potential benefits and limitations. It is important to note that WBV may not be suitable for all individuals with PFPS.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) can significantly affect an individual's ability perform to functional activities, such as walking, running, climbing stairs, and sitting for prolonged periods.

PFPS is often associated with pain and discomfort in the front of the knee, which can limit an individual's range of motion and cause difficulty with weight-bearing activities. The pain may also be exacerbated by activities that involve bending the knee, such as squatting or kneeling.

Whole body vibration (WBV) has been suggested as a potential intervention for patellofemoral pain syndrome (PFPS). Some studies have shown that WBV can improve muscle strength, balance, and proprioception, which are all factors that may contribute to PFPS. Additionally, WBV may help reduce pain and improve functional abilities in individuals with PFPS.

However, the evidence for the effectiveness of WBV as an intervention for PFPS is still limited, and more research is needed to fully understand its potential benefits and limitations. It is important to note that WBV may not be suitable for all individuals with PFPS.

HYPOTHESES:

There will be no significant difference on dorsi/planter flexor ratio , functional activities and pain level after adding the whole body vibration to traditional treatment of PFPS

RESEARCH QUESTION:

What is the impact of whole-body vibration on dorsi/planter flexor ratio, functional activities and pain levels in individuals with PFPS?

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults aged 18 -35 years
2. Symptoms: Pain in the anterior or retro patellar knee region during activities such as running, jumping, squatting, or prolonged sitting
3. Duration: Pain lasting at least 6 weeks

Exclusion Criteria:

1. Presence of other knee conditions: Individuals with PFPS who also have other knee conditions such as ligament or meniscal injuries, osteoarthritis, or patellar tendinopathy may be excluded.
2. History of knee surgery: Patients who have undergone any knee surgery may be excluded as this may affect the outcomes of the study.
3. Systemic conditions: Patients with systemic conditions that may affect the musculoskeletal system such as rheumatoid arthritis or lupus may be excluded.
4. Pregnancy: Pregnant women with PFPS may be excluded as pregnancy may affect the outcomes of the study.
5. Inability to comply with study requirements: Patients who are unable to comply with the study requirements such as attending follow-up appointments or completing questionnaires may be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Dorsi/planter torque ratio | one month
  dorsi/planter torque ratio will be measured through the Biodex System 4-Pro Isokinetic Strength Dynamometer for assessment of muscle torque
functional activities | one month
  Kujala Anterior Knee Pain Scale, which includes questions related to functional activities.
Pain intensity | one month
  10 cm Visual Analogue Scale (VAS) was used to assess pain intensity during activity in patients with patellofemoral pain (PFP). The scale ranged from 0, indicating "no pain," to 100, representing the "worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy , cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: study protocol